CLINICAL TRIAL: NCT05767905
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 3-PERIOD, CROSSOVER, SINGLE-DOSE, 2-PART STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE EFFECT OF TABLET FORMULATION AND FOOD ON THE RELATIVE BIOAVAILABILITY OF PF-06821497
Brief Title: A Study to Understand the Effect of Tablet Formulation and Food on PF-06821497 in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C2321005; NCT05767905 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: PF-06821497; Relative Bioavailability; Food Effect

STUDY DESIGN:
Masking Description: Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: PF-06821497 Sequence 1 (Experimental): Participants randomized to Sequence 1 will receive Treatments A, B, and C in Periods 1 through 3, respectively in the form of tablets by mouth.
  Interventions:
  * Drug: Single dose of PF-06821497 Treatment A
  * Drug: Single dose of PF-06821497 Treatment B
  * Drug: Single dose of PF-06821497 Treatment C
  Interventions: Drug: PF-06821497 Treatment A; Drug: PF-06821497 Treatment B; Drug: PF-06821497 Treatment C
- Part 1: PF-06821497 Sequence 2 (Experimental): Participants randomized to Sequence 2 will receive Treatments B, A and C in Periods 1 through 3, respectively in the form of tablets by mouth.
  Interventions:
  * Drug: Single dose of PF-06821497 Treatment A
  * Drug: Single dose of PF-06821497 Treatment B
  * Drug: Single dose of PF-06821497 Treatment C
  Interventions: Drug: PF-06821497 Treatment A; Drug: PF-06821497 Treatment B; Drug: PF-06821497 Treatment C
- Part 2: PF-06821497 Sequence 1 (Experimental): Participants randomized to Sequence 1 will receive Treatments D, E and F in Periods 1 through 3, respectively in the form of tablets by mouth.
  Interventions:
  * Drug: Single dose of PF-06821497 Treatment D
  * Drug: Single dose of PF-06821497 Treatment E
  * Drug: Single dose of PF-06821497 Treatment F
  Interventions: Drug: PF-06821497 Treatment D; Drug: PF-06821497 Treatment E; Drug: PF-06821497 Treatment F

INTERVENTIONS:
Drug: PF-06821497 Treatment A — A single dose of PF-06821497 administered under fasting conditions.
  Arms: Part 1: PF-06821497 Sequence 1; Part 1: PF-06821497 Sequence 2
Drug: PF-06821497 Treatment B — A single dose of PF-06821497 administered under fasting conditions.
  Arms: Part 1: PF-06821497 Sequence 1; Part 1: PF-06821497 Sequence 2
Drug: PF-06821497 Treatment C — A single dose of PF-06821497 administered under fasting conditions.
  Arms: Part 1: PF-06821497 Sequence 1; Part 1: PF-06821497 Sequence 2
Drug: PF-06821497 Treatment D — A single dose of PF-06821497 administered under fasting conditions.
  Arms: Part 2: PF-06821497 Sequence 1
Drug: PF-06821497 Treatment E — A single dose of PF-06821497 administered after low fat meal
  Arms: Part 2: PF-06821497 Sequence 1
Drug: PF-06821497 Treatment F — A single dose of PF-06821497 administered after high fat meal.
  Arms: Part 2: PF-06821497 Sequence 1

SUMMARY:
The purpose of this study is to understand the effect of tablet formulation and presence of food on the study medicine PF-06821497 in healthy adult participants.

The study is seeking for male and female participants who:

* Are 18 years of age or more.
* Are confirmed to be healthy after performing some medical and physical tests.
* Weigh more than 50kgs of body weight and have a body mass index of 17 and a half kg per meter squared or more.

The study consists of two parts. In each part of the study, the selected participants will take part in 3 study periods to receive 3 different treatments which are randomly assigned. There will also be a 5-day gap between each study period. This is done so that the medicine is passed out of the body before the start of next study period.

Each treatment consists of a single dose of PF-06821497. The treatments differ by tablet formulation and/or whether the medicine is to be given with food or without food conditions.

How the medicine is processed in the body will be studied after giving the medicines to the participants. This will be done by collecting blood samples after each administration. The results will be used to see the effect of tablet formulation and presence of food on the amount of PF-06821497 available in the blood of the participants.

In each part, participants will be on the study up to 10 weeks, including the screening and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age, inclusive, at screening.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECGs.
* BMI of ≥17.5 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) or prior allergic reaction to any component of PF-06821497.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants (12 participants in Part 1 and 6 participants in Part 2) were randomized and assigned to study treatments.
Groups:
- Part 1: PF-06821497 Form 1 250 mg -> PF-06821497 Form 2 250 mg -> PF-06821497 Form 3 250 mg.: Participants received PF-06821497 (formulation 1) 250 mg material sparing tablet (MST) on Day 1 of period 1 under fasted condition, and after a minimum of 5-day washout period, participants received PF-06821497 (formulation 2) 250 mg wet granulation (WG) tablet on Day 1 of period 2 under fasted condition. Then after a minimum of 5-day washout period, participants received PF-06821497 (formulation 3) 250 mg WG tablet (larger API particle size) on Day 1 of period 3 under fasted condition.
- Part 1: PF-06821497 Form 2 250 mg -> PF-06821497 Form 1 250 mg -> PF-06821497 Form 3 250 mg: Participants received PF-06821497 (formulation 2) 250 mg WG tablet on Day 1 of period 1 under fasted condition, and after a minimum of 5-day washout period, participants received PF-06821497 (formulation 1) 250 mg MST tablet on Day 1 of period 2 under fasted condition. Then after a minimum of 5-day washout period, participants received PF-06821497 (formulation 3) 250 mg WG tablet (larger API particle size) on Day 1 of period 3 under fasted condition.
- Part 2:PF-06821497 1250 mg Fasted >PF-06821497 1250 mg Fed Low-fat >PF-06821497 1250 mg Fed High-fat: Participants received PF-06821497 (formulation 2) 1250 mg WG tablet on Day 1 of period 1 under fasted condition, and after a minimum of 5-day washout period, participants received a received a low-fat, low-calorie breakfast 30 minutes prior to dosing of PF-06821497 (formulation 2) 1250 mg WG tablet on Day 1 of period 2. Then after a minimum of 5-day washout period, participants received a a high-fat, high-calorie breakfast 30 minutes prior to dosing of PF-06821497 (formulation 2) 1250mg WG tablet.
Period: Overall Study
Arm/Group | Part 1: PF-06821497 Form 1 250 mg -> PF-06821497 Form 2 250 mg -> PF-06821497 Form 3 250 mg. | Part 1: PF-06821497 Form 2 250 mg -> PF-06821497 Form 1 250 mg -> PF-06821497 Form 3 250 mg | Part 2:PF-06821497 1250 mg Fasted >PF-06821497 1250 mg Fed Low-fat >PF-06821497 1250 mg Fed High-fat
Started | 6 | 6 | 6
Completed | 6 | 6 | 5
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study, and the results were presented by part.
Groups:
- Part 1: In Part 1, each enrolled participant participated in 3 study periods to receive 3 different treatments(Treatment A: Single 250 mg dose (1 × 250 mg) of MST tablet formulation (Formulation 1), fasted; Treatment B: Single 250 mg dose (1 × 250 mg) of WG tablet formulation (Formulation 2), fasted; Treatment C: Single 250 mg dose (1 × 250 mg) of WG tablet formulation (larger API particle size) (Formulation 3), fasted.) according to the sequence determined by randomization with 5-day washouts between PF-06821497 administration.
- Part 2: In Part 2, each enrolled participant participated in 3 study periods to receive 3 different treatments (Treatment D: Single 1250 mg dose (5 × 250 mg) of WG tablet formulation (Formulation 2), fasted; Treatment E: Single 1250 mg dose (5 × 250 mg) of WG tablet formulation (Formulation 2), fed, low-fat; Treatment F: Single 1250 mg dose (5 × 250 mg) of WG tablet formulation (Formulation 2), fed, high-fat.) according to the sequence determined by randomization with 5-day washouts between PF-06821497 administration.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Customized [Count of Participants; unit: Participants]
  18 -44 years | 7 | 2 | 9
  45 - 64 years | 4 | 3 | 7
  >= 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 4 | 11
  Black or African American | 3 | 1 | 4
  Black or African American, White | 1 | 0 | 1
  Black or African American, White, American Indian or Alaska Native | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06821497
Description: The AUCinf was determined by AUClast + (Clast/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. AUClast is the area under the concentration-time curve from 0 to time of last measurable concentration
Time Frame: Days 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose), 2 and 3 in Periods 1 to 3.
Population: The pharmacokinetic (PK) parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PF-06821497 PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 1 PF-06821497 Form 1 250 mg Fasted: Following an overnight fast of at least 10 hours, and after the collection of the pre-dose PF-06821497 PK sample on Day 1 of each period, participants received a 250 mg dose of PF-06821497 material sparing tablet (MST).
- Part 1 PF-06821497 Form 2 250 mg Fasted: Following an overnight fast of at least 10 hours, and after the collection of the pre-dose PF-06821497 PK sample on Day 1 of each period, participants received a 250 mg dose of PF-06821497 wet granulation (WG) tablet.
- Part 1 PF-06821497 Form 3 250 mg Fasted: Following an overnight fast of at least 10 hours, and after the collection of the pre-dose PF-06821497 PK sample on Day 1 of each period, participants received a 250 mg dose of PF-06821497 WG tablet (larger API particle size).
- Part 2 PF-06821497 Form 2 1250 mg Fasted: Following an overnight fast of at least 10 hours, and after the collection of the pre-dose PF-06821497 PK sample on Day 1, participants received a 1250 mg dose of PF-06821497 WG tablet.
- Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat: Following an overnight fast of at least 10 hours and after the collection of pre-dose PF-06821497 PK sample on Day 1, participants received a low-fat, low-calorie breakfast 30 minutes prior to a dose of PF-06821497 1250mg WG tablet
- Part 2 PF-06821497 Form 2 1250 mg Fed High-fat: Following an overnight fast of at least 10 hours and after the collection of pre-dose PF-06821497 PK sample on Day 1, participants received a high-fat, high-calorie breakfast 30 minutes prior to a dose of PF-06821497 1250mg WG tablet
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 6 | 5
ng*hr/mL | 3302 (33) | 3375 (29) | 3479 (39) | 11220 (48) | 22810 (24) | 25690 (35)
Statistical Analysis 1: Comparison: Part 1 PF-06821497 Form 1 250 mg Fasted vs Part 1 PF-06821497 Form 3 250 mg Fasted; Part 1 PF-06821497 Form 1 250 mg Fasted was the Reference treatment and Part 1 PF-06821497 Form 3 250 mg Fasted was the Test treatment; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain: 1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 108.49, 90% CI 2-sided [100.55 to 117.05]
Statistical Analysis 2: Comparison: Part 1 PF-06821497 Form 2 250 mg Fasted vs Part 1 PF-06821497 Form 3 250 mg Fasted; Part 1 PF-06821497 Form 3 250 mg Fasted was the Test treatment and Part 1 PF-06821497 Form 2 250 mg Fasted was the Reference treatment; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 106.16, 90% CI 2-sided [98.39 to 114.54]
Statistical Analysis 3: Comparison: Part 2 PF-06821497 Form 2 1250 mg Fasted vs Part 2 PF-06821497 Form 2 1250 mg Fed High-fat; Part 2 PF-06821497 Form 2 1250 mg Fed High-fat was the Test treatment and Part 2 PF-06821497 Form 2 1250 mg Fasted was the Reference treatment; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 228.99, 90% CI 2-sided [178.67 to 293.48]
Statistical Analysis 4: Comparison: Part 2 PF-06821497 Form 2 1250 mg Fasted vs Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat; Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat was the Test treatment and Part 2 PF-06821497 Form 2 1250 mg Fasted was the Reference treatment; Test type: Other; ratio = 207.19, 90% CI 2-sided [164.41 to 261.09]
Statistical Analysis 5: Comparison: Part 1 PF-06821497 Form 1 250 mg Fasted vs Part 1 PF-06821497 Form 2 250 mg Fasted; Part 1 PF-06821497 Form 1 250 mg Fasted was the Reference treatment, and Part 1 PF-06821497 Form 2 250 mg Fasted was the Test treatment; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 102.19, 90% CI 2-sided [95.55 to 109.30]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for PF-06821497.
Description: The Cmax was observed directly from data.
Time Frame: Days 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose), 2 and 3 in Periods 1 to 3.
Population: The PK concentration population was defined as all participants randomized and treated who had at least 1 PF-06821497 concentration in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 6 | 5
ng/mL | 862.6 (50) | 1023 (35) | 1255 (37) | 2699 (31) | 7685 (28) | 8905 (7)
Statistical Analysis 1: Comparison: Part 1 PF-06821497 Form 1 250 mg Fasted vs Part 1 PF-06821497 Form 3 250 mg Fasted; Part 1 PF-06821497 Form 3 250 mg Fasted was the Test treatment and Part 1 PF-06821497 Form 1 250 mg Fasted was the Reference treatment; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 145.49, 90% CI 2-sided [121.29 to 174.53]
Statistical Analysis 2: Comparison: Part 1 PF-06821497 Form 2 250 mg Fasted vs Part 1 PF-06821497 Form 3 250 mg Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 122.64, 90% CI 2-sided [102.24 to 147.12]
Statistical Analysis 3: Comparison: Part 2 PF-06821497 Form 2 1250 mg Fasted vs Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat; [analysis description as in outcome 1, analysis 4]; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 284.72, 90% CI 2-sided [226.39 to 358.06]
Statistical Analysis 4: Comparison: Part 2 PF-06821497 Form 2 1250 mg Fasted vs Part 2 PF-06821497 Form 2 1250 mg Fed High-fat; [analysis description as in outcome 1, analysis 3]; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 327.87, 90% CI 2-sided [256.90 to 418.44]
Statistical Analysis 5: Comparison: Part 1 PF-06821497 Form 1 250 mg Fasted vs Part 1 PF-06821497 Form 2 250 mg Fasted; [analysis description as in outcome 1, analysis 5]; Test type: Other; Mixed Models Analysis; Mixed Model was fitted to obtain:1.Ratio of geometric means 2.90% CI of ratio of geometric means; ratio = 118.63, 90% CI 2-sided [96.36 to 146.06]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs).
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, was considered serious.
Time Frame: From screening up to Day 35
Population: The safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants was analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 6 | 5
Participants | 5 | 4 | 2 | 3 | 3 | 2

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Safety laboratory assessments included urinalysis, hematology, chemistry and other. All the safety laboratory samples were collected following at least a 4-hour fast.
Time Frame: From screening up to Day 3 of Period 3, and prior to early termination/discontinuation, up to 10 weeks.
Population: The analysis population included all participants randomly assigned to study intervention and who took at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 PF-06821497 Form 2 1250 mg Fasted: Following an overnight fast of at least 10 hours, and after the collection of the pre-dose PF-06821497 PK sample on Day 1 of each period, participants received a 250 mg dose of PF-06821497 WG tablet (larger API particle size).
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 1 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant ECG Findings
Description: Single 12-lead electrocardiogram or electrocardiography (ECG) readings were taken at approximately each test. All ECG assessments were made after at least a 5-minute rest in a supine position and prior to any blood draws or vital sign measurements.
Time Frame: From screening up to Day 3 of Period 3, and prior to early termination/discontinuation, up to 10 weeks.
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 6 | 5
Participants
  PR Interval, aggregate (msec), value > = 300 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, aggregate (msec), %Change >= 25/50% | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration, aggregate (msec), value >= 140 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration, aggregate (msec), %Change >= 50% | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval, aggregate (msec), value >= 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval, aggregate (msec), 450 <= value < 480 | 0 | 1 | 0 | 0 | 0 | 0
  QTcB Interval, aggregate (msec), 480 <= value < 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval, aggregate (msec), value >= 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval, aggregate (msec), 30 <= change < 60 | 0 | 0 | 1 | 0 | 0 | 0
  QTcB Interval, aggregate (msec), change >= 60 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, aggregate (msec), 450 <= value < 480 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, aggregate (msec), 480 <= value < 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, aggregate (msec), value >= 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, aggregate (msec), 30 <= change < 60 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, aggregate (msec), change >= 60 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to Day 35.
Description: Serious adverse events(SAE) and non-serious AEs were recorded on the case report form.
Arm/Group | Part 1 PF-06821497 Form 1 250 mg Fasted | Part 1 PF-06821497 Form 2 250 mg Fasted | Part 1 PF-06821497 Form 3 250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fasted | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/6 | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12 | 2/12 | 3/6 | 3/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 PF-06821497 Form 1 250 mg Fasted (N=12) | Part 1 PF-06821497 Form 2 250 mg Fasted (N=12) | Part 1 PF-06821497 Form 3 250 mg Fasted (N=12) | Part 2 PF-06821497 Form 2 1250 mg Fasted (N=6) | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat (N=6) | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat (N=5)
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 PF-06821497 Form 1 250 mg Fasted (N=12) | Part 1 PF-06821497 Form 2 250 mg Fasted (N=12) | Part 1 PF-06821497 Form 3 250 mg Fasted (N=12) | Part 2 PF-06821497 Form 2 1250 mg Fasted (N=6) | Part 2 PF-06821497 Form 2 1250 mg Fed Low-fat (N=6) | Part 2 PF-06821497 Form 2 1250 mg Fed High-fat (N=5)
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Nail avulsion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05767905/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT05767905/SAP_001.pdf